CLINICAL TRIAL: NCT03954067
Title: A Phase 1, Open-label Study of ASP9801, an Oncolytic Virus, Administered by Intratumoral Injection as a Single Agent and in Combination With Pembrolizumab in Subjects With Advanced/Metastatic Solid Tumors
Brief Title: A Study of an Intratumoral Oncolytic Virus in Patients With Advanced Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 9801-CL-0101; KEYNOTE-B26 (Other: Merck Sharp & Dohme Corp); MK-3475-B26 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2019-05-14; First posted 2019-05-17 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Cancer; Solid Tumors; Advanced Cancer
Keywords: immunotherapy; vaccinia virus; visceral lesions; cutaneous lesions; intratumoral injection; ASP9801; subcutaneous lesions; oncolytic virus
MeSH Terms: conditions — Neoplasm Metastasis; Vaccinia | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Dose Escalation - cutaneous or subcutaneous lesions (Experimental): Participants will receive ASP9801 (1x10^7 pfu/mL) on days 1 and 15 of 28 day cycles to determine the recommended phase 2 dose. After cycle 2, participants who have not met any discontinuation criteria and receiving clinical benefit may be treated on continuous cycles until treatment discontinuation criteria are met.
  Interventions: Biological: ASP9801
- Dose Escalation - visceral lesions (Experimental): Participants will receive ASP9801 (1x10^8 pfu/mL) on days 1 and 15 of 28 day cycles to determine the recommended phase 2 dose. After cycle 2, participants who have not met any discontinuation criteria and receiving clinical benefit may be treated on continuous cycles until treatment discontinuation criteria are met.
  Interventions: Biological: ASP9801
- Dose Expansion (Monotherapy) - cutaneous or subcutaneous lesions (Experimental): Participants will receive ASP9801 (1x10^8 pfu/mL) on days 1 and 15 of 28 day cycles at the dose recommended by the dose escalation phase. After cycle 2, participants who have not met any discontinuation criteria and receiving clinical benefit may be treated on continuous cycles until treatment discontinuation criteria are met.
  Interventions: Biological: ASP9801
- Dose Expansion (Monotherapy) - visceral lesions (Experimental): Participants will receive ASP9801 (5x10^8 pfu/mL) on days 1 and 15 of 28 day cycles at the dose recommended by the dose escalation phase. After cycle 2, participants who have not met any discontinuation criteria and receiving clinical benefit may be treated on continuous cycles until treatment discontinuation criteria are met.
  Interventions: Biological: ASP9801
- Dose Expansion (Monotherapy Induction) - cutaneous or subcutaneous lesions (Experimental): Participants will receive ASP9801 (5x10^8 pfu/mL) on days 1, 8, 15 and 22 of the first 28 day cycle. Participants will receive ASP9801 on days 1 and 15 on the second 28 day cycle at the dose recommended by the dose escalation phase. After cycle 2, participants who have not met any discontinuation criteria and receiving clinical benefit may be treated on continuous cycles until treatment discontinuation criteria are met.
  Interventions: Biological: ASP9801
- Dose Expansion (Combination Therapy) - cutaneous or subcutaneous lesions (Experimental): Participants will receive ASP9801 (1x10^8 pfu/mL) on days 1 and 15 of 28 day cycles at the dose recommended by the dose escalation phase. Participants will also receive pembrolizumab starting on day 1 and once every 6 weeks. After cycle 2, participants who have not met any discontinuation criteria and receiving clinical benefit may be treated on continuous cycles until treatment discontinuation criteria are met.
  Interventions: Combination Product: Pembrolizumab
- Dose Expansion (Combination Induction Therapy) - cutaneous or subcutaneous lesions (Experimental): Participants will receive ASP9801 (5x10^8 pfu/mL) on days 1, 8, 15 and 22 of first 28 day cycle at the dose recommended by the dose escalation phase. Participants will also receive pembrolizumab starting on day 1 and once every 6 weeks. Participants will receive ASP9801 on days 1 and 15 on the second 28 day cycle at the dose recommended by the dose escalation phase. After cycle 2, participants who have not met any discontinuation criteria and receiving clinical benefit may be treated on continuous cycles until treatment discontinuation criteria are met.
  Interventions: Combination Product: Pembrolizumab
- Dose Expansion (Combination Therapy) - visceral lesions (Experimental): Participants will receive ASP9801 (5x10^8 pfu/mL) on days 1 and 15 of 28 day cycles at the dose recommended by the dose escalation phase. Participants will also receive pembrolizumab starting on day 1 and once every 6 weeks. After cycle 2, participants who have not met any discontinuation criteria and receiving clinical benefit may be treated on continuous cycles until treatment discontinuation criteria are met.
  Interventions: Combination Product: Pembrolizumab

INTERVENTIONS:
Biological: ASP9801 — Administered by intratumoral injection
  Arms: Dose Escalation - cutaneous or subcutaneous lesions; Dose Escalation - visceral lesions; Dose Expansion (Monotherapy Induction) - cutaneous or subcutaneous lesions; Dose Expansion (Monotherapy) - cutaneous or subcutaneous lesions; Dose Expansion (Monotherapy) - visceral lesions
Combination Product: Pembrolizumab — Administered by Intravenous Infusion
  Other Names: KEYTRUDA®
  Arms: Dose Expansion (Combination Induction Therapy) - cutaneous or subcutaneous lesions; Dose Expansion (Combination Therapy) - cutaneous or subcutaneous lesions; Dose Expansion (Combination Therapy) - visceral lesions

SUMMARY:
The purpose of this study is to assess the safety and tolerability of ASP9801 and to determine the recommended phase 2 dose (RP2D). The study will also evaluate antitumor activity, objective response rate, pharmacokinetics and virus shedding of ASP9801 as a single agent, as well as in combination with pembrolizumab, an anti-programmed cell death protein 1 (PD-1) checkpoint inhibitor.

DETAILED DESCRIPTION:
The study consists of two parts: dose escalation and recommended phase 2 dose expansion. Each part of the study will include two separate groups of participants. Group A will include participants who will have cutaneous/subcutaneous tumors injected, and group B will include participants who will have visceral tumors injected. In dose escalation part only ASP9801 will be assessed. In dose expansion part along with ASP9801 (monotherapy) ASP9801 + Pembrolizumab (combination therapy) will be assessed. The study will consist of the following periods: screening, initial treatment period (two 28 day cycles), optional extended treatment period (continued 28 day cycles) and a follow up period (safety and survival follow up).

ELIGIBILITY:
Inclusion Criteria:

* Subject must have histologically- or cytologically-confirmed diagnosis of advanced or metastatic solid tumor(s).
* Subject has measurable disease as determined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. At least 1 lesion must be suitable for intratumoral (IT) injection. Lesions for injection must be ≥ 10 mm and ≤ 60 mm in longest diameter.
* Subject has had disease progression after, been intolerant to, or has refused all available therapies that are known to confer clinical benefit. Note: There is no limit to the number of prior treatment regimens.
* Subject has a predicted life expectancy ≥ 12 weeks.
* Subject has at least 2 sites of disease suitable for biopsy and is willing and able to undergo required tumor biopsies according to the treating institution's guidelines at screening and during study treatment.
* Subject has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* A female subject is eligible to participate if she is not pregnant as documented by negative pregnancy test within 72 hours prior to treatment and at least 1 of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) OR
  * WOCBP who agrees to follow the contraceptive guidance throughout the treatment period and for at least 180 days after the final study investigational product (IP) administration.
* Female subject must agree not to breastfeed starting at screening, and throughout the study period and 180 days after the final study IP administration.
* Female subject must not donate ova starting at screening, and throughout the study period and for 180 days after the final study IP administration.
* Male subject must agree to remain abstinent or use a condom throughout the study period and for 180 days after the final study IP administration.
* Male subject with female partner(s) of childbearing potential must agree to use contraception during the treatment period and for at least 180 days after the final study IP administration.
* Male subject must not donate sperm during the treatment period and for at least 180 days after the final study IP administration.
* Subject must be willing and able to comply with the study requirements including prohibited concomitant medication restrictions.
* Subject agrees not to participate in another interventional study while receiving study IP.
* Subject has the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Subject has ongoing toxicity ≥ National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE) grade 2 attributable to prior antineoplastic therapies considered clinically significant.
* Subject who has had major surgery ≤ 4 weeks of screening. Subjects must have recovered from prior procedures and/or any complications from surgery prior to starting study treatment.
* Subject is concurrently participating in another interventional study or has received an investigational product ≤ 30 days or 5 half-lives whichever is shorter, prior to first IP administration.
* Subject with symptomatic or untreated central nervous system (CNS) metastases or leptomeningeal disease. Subjects with treated symptomatic brain metastases should be neurologically stable (without evidence of progression by imaging for at least 4 weeks prior to screening and any neurologic symptoms have returned to baseline) and off steroids for at least 2 weeks prior to first IP administration. Subjects with carcinomatous meningitis are excluded regardless of clinical stability.
* Subject with active or prior autoimmune or inflammatory disorders requiring systemic therapy within past 2 years (including inflammatory skin conditions or severe eczema, inflammatory bowel disease (e.g., colitis or Crohn's disease), diverticulitis (with the exception of diverticulosis), celiac disease, systemic lupus erythematosus, Sarcoidosis syndrome, Wegener syndrome (granulomatosis with polyangiitis), Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.

The following are exceptions to this criterion:

* Subject with vitiligo or alopecia
* Subject with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
* Any chronic skin condition that does not require systemic therapy

  * Subject with another malignancy that currently requires treatment.
  * Subject with only tumors encasing major vascular structures such as the carotid artery, tumors adjacent to vital neurovascular structures or tumors in locations that are at high risk for adverse events (AEs) or otherwise not considered appropriate for IT injection. Subjects with such tumors that have other injectable tumors would be eligible.
  * Subject with inadequate organ and marrow functions meeting any of the below criteria:
* Leukocytes < 3000/μL
* Absolute neutrophil count < 1500/μL
* Platelets < 100,000/μL
* Hemoglobin (Hgb) < 9 g/dL (Criteria must be met without packed red blood cell transfusion within the prior 2 weeks. Subjects can be on stable dose of erythropoietin [≥ approximately 3 months])
* International normalized ratio (INR) > 1.5 × ULN and/or activated partial thromboplastin time (aPTT) > 1.5 × institutional normal limits, except for subjects in Group B (Visceral Lesions) escalation and expansion groups where INR and aPTT must be normal
* Total Bilirubin (TBL) > 1.5 × institutional normal limits (subjects with known Gilbert syndrome who are excluded if TBL > 3.0 × institutional normal limits or direct bilirubin > 1.5 × institutional normal limits)
* Aspartate aminotransferase (AST) and Alanine transaminase (ALT) > 2.5 × institutional normal limits. Subjects with tumors in the liver AST and ALT > 5 × institutional normal limits.
* Albumin < 3.0 g/dL
* Creatinine > 1.5 × institutional normal limits

  * Subject with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of first administration of study IP. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
  * Subject has an uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, any form of substance abuse or psychiatric illness/social situations that would limit compliance with study visits or requirements or a condition that could invalidate communication with the investigator.
  * Subject is positive for human immunodeficiency virus, hepatitis B surface antigen, hepatitis B core immunoglobulin or immunoglobulin G (IgG) antibody or hepatitis C (IgG or ribonucleic acid (RNA) test) indicating acute or chronic infection.
  * Subject has a history of moderate to severe ascites, clinically significant and/or rapidly accumulating ascites, bleeding esophageal varices, hepatic encephalopathy or pericardial and/or pleural effusions related to liver insufficiency within 6 months of screening. Mild ascites that does not preclude safe IT injection of ASP9801 is allowed.
  * Subject has a clinically significant abnormal electrocardiogram (ECG) at screening.
  * Subject has symptomatic cardiovascular disease within the preceding 12 months unless cardiology consultation and clearance has been obtained for study participation, including but not limited to the following: significant coronary artery disease (e.g., requiring angioplasty or stenting), acute myocardial infarction or unstable angina pectoris < 3 months prior to screening, uncontrolled hypertension, clinically significant arrhythmia or congestive heart failure (New York Heart Association grade ≥ 2).
  * Subject has medical conditions that predispose the subject to untoward medical risk in the event of volume loading (e.g., intravenous fluid bolus infusion), tachycardia or hypotension during or following treatment with ASP9801.
  * Subject has a known or suspected hypersensitivity to ASP9801 or any components of the formulation used, including prior adverse reaction to vaccinia (e.g., as smallpox vaccine).
  * Subject has had previous exposure with ASP9801.
  * Subject has an active infection requiring systemic therapy.
  * Subject with known history of active Bacillus Tuberculosis.
  * Subject has received prior therapy with an anti-PD-1, anti-programmed cell death ligand 1 (PD-L1), or anti-programmed cell death ligand 2 (PD-L2) agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., cytotoxic T-lymphocyte-associated protein 4, OX 40, CD137) and was discontinued from that treatment due to an immune-related adverse event.
  * Subject has received prior radiation therapy within 2 weeks of start of study treatment. Subject must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤ 2 weeks of radiotherapy) to non-CNS disease.
  * Subject has received a live vaccine within 30 days prior to the first dose of study drug.

Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, bacillus Calmette-Guérin and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.

* Subject has severe hypersensitivity (≥ grade 3) to pembrolizumab and/or any of its excipients, or history of ≥ grade 2 infusion reactions that were not prevented by adequate premedication.
* Subject has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Subject has had an allogeneic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) - dose escalation part | Up to 28 days
  Incidence of dose limiting toxicities
Safety and tolerability assessed by Adverse Events (AEs) | Up to 12 months
  An AE is any untoward medical occurrence in a subject administered an investigational product (IP), and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IP whether or not considered related to the IP.
Number of participants with laboratory value abnormalities and/or adverse events | Up to 12 months
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities and /or adverse events | Up to 12 months
  Number of participants with potentially clinically significant vital sign values.
Safety assessed by 12- lead electrocardiograms (ECGs) adverse events | Up to 12 months
  12-lead ECGs will be read and assessed locally. Any clinically significant adverse changes on the ECG will be reported as Adverse Events.

SECONDARY OUTCOMES:
Percent change from baseline in antitumor activity of ASP9801 | Up to 12 months
  Percent change from baseline in sum of diameters of injected tumors per Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1 and immune modified response evaluation criteria in solid tumors (imRECIST)
Objective Response Rate per imRECIST | Up to 12 months
  Partial Response (PR) + Complete Response (CR) per imRECIST
ASP9801 viral DNA in blood | Up to 12 months
  Viral DNA load will be summarized by cohort using descriptive statistics.
Viral shedding of ASP9801 in saliva | Up to 12 months
  Viral DNA will be analyzed by quantitative polymerase chain reaction (qPCR).
Viral shedding of ASP9801 in urine | Up to 12 months
  Viral DNA will be analyzed by qPCR.
Viral shedding of ASP9801 in skin (cutaneous/subcutaneous only) | Up to 12 months
  Viral DNA will be analyzed by qPCR.
Objective Response Rate per Response Evaluation Criteria in Solid Tumors version (RECIST) 1.1 | Up to 12 months
  Partial Response (PR) + Complete Response (CR) per RECIST 1.1.
Change in Programmed Cell Death Ligand 1 (PD-L1) Expression in Tumor | Up to 12 months
  Changes in level of PDL1 expression in tumors will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (17):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arizona - Arizona Cancer Center, Tucson, Arizona
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - The University of Chicago Medical Center, Chicago, Illinois
  - University of Kentucky, Markey Cancer Center, Lexington, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Roswell Park Cancer Institute - Medical Oncology, Buffalo, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - The University of Texas - MD Anderson Cancer Center, Houston, Texas
  - UVA Cancer Center, Charlottesville, Virginia
  - VCU Massey Cancer Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/9801-CL-0101/
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=14539&tenant=MT_AST_9011